CLINICAL TRIAL: NCT06016348
Title: Predictors of Good Outcomes in Thrombectomy for Stroke Patients Within 24 Hours From Symptom Onset With Large Infarct Core
Brief Title: PROMISE: PRedictors Of Good outcoMes in Thrombectomy for Large Infarct Core Stroke Evaluation
Status: Completed | Type: Observational
Sponsor: 115 People's Hospital (Other Government)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Trung Nguyen, Principal Investigator, 115 People's Hospital
Other Study IDs: 115
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: large core; Low ASPECTS; Endovascular treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good outcome: mRS of 0-3; mRS of 0-2
  Interventions: Procedure: Endovascular treatment
- Unfavorable outcomes: mRS of 4-6
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Procedure: Endovascular treatment — This procedure is instrumental in restoring cerebral blood flow by addressing the clot-induced obstruction within brain-supplying blood vessels.
  Other Names: Mechanical thrombectomy

SUMMARY:
Identify the factors associated with a favorable clinical outcome in participants with acute ischemic stroke and large core infarcts within 24 hours of onset who are treated with endovascular intervention.

DETAILED DESCRIPTION:
In 2022 and early 2023, three randomized controlled trials-RESCUE-JAPAN LIMIT, SELECT 2, and ANGEL ASPECT-were published in the New England Journal of Medicine. These trials demonstrated the effectiveness and safety of endovascular intervention using clot retrieval devices in participants with acute ischemic stroke and large core infarcts. However, the rate of participants achieving a good recovery remains low, while the mortality and disability rates are very high.

Moreover, in Vietnam, the acute stroke treatment process has not been optimized, and the facilities and equipment for monitoring neurointensive care are not fully equipped. As a result, endovascular intervention using clot retrieval devices in participants with large core infarcts has not been widely implemented in the investigator's country, and the effectiveness and safety of this treatment method have not been clearly evaluated.

Addressing this issue is crucial for improving the quality of life and reducing the mortality and disability rates caused by stroke in this participant group. This study aims to provide new insights into the use of endovascular intervention for treating acute ischemic stroke with a large core infarct volume, thereby supporting clinical decision-making and improving treatment outcomes for participants with acute ischemic stroke and large core infarcts.

We hypothesize that core infarction is not the sole factor for excluding patients from potent thrombectomy therapy. We aim to determine predictors of favorable and unfavorable outcomes following thrombectomy in patients with large core strokes. Secondly, we aim to build a multivariable calculator to predict good or poor outcomes after thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-year-old
* Patients presenting with acute ischaemic stroke within 24 hours of stroke onset
* Received mechanical thrombectomy within 24 hours of stroke onset
* Imaging criteria include:

  * Large vessel occlusion on CT Angiography or MR Angiography (MRA) including tandem occlusion of the internal carotid artery and middle cerebral artery or internal carotid artery.
  * Core infarct criteria:

    1. ASPECTS ≤5 on non-contrast CT or diffusion-weighted imaging (DWI).
    2. ASPECTS score >5 and core infarct volume of 50-150 ml on CT perfusion (CTP) or reduced cerebral blood flow (rCBF) <30% on CTP or apparent diffusion coefficient (ADC) <620 × 10-6 mm2/s on DWI.

Exclusion Criteria:

* Patients presenting with acute ischaemic stroke >24 hours of stroke onset
* Intracranial hemorrhage identified by CT or MRI
* Pre-stroke modified Rankin Score (mRS) score of >2 (indicating previous disability)
* Any terminal illness such that the patient has a life expectancy of less than 1 year.
* Patients with active cancer and undergoing treatment for cancer are excluded,
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All adult patients underwent mechanical thrombectomy within 24 hours from symptom onset.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
The Modified Rankin Scale (mRS) of 0-3 | 90 (± 14 days) after procedure
  The rate of independent ambulation (mRS 0-3). The scale runs from 0-6, running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
mRS of 0-2 | 90 (± 14 days) after procedure
  The rate of functional independence (mRS 0-2)
mRS of 0-5 | 90 (± 14 days) after procedure
  The survival rate
Symptomatic intracerebral hemorrhage (sICH) | 72 hours
  sICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 72 hours or any hemorrhage leading to death.
Early neurological deterioration | 72 hours
  Clinical worsening that was higher by ≥4 points than the value at baseline during the first 72 h after ischaemic stroke.

CONTACTS AND LOCATIONS:
Locations (4):
- Vietnam (4):
  - Can Tho Central General Hospital, Can Tho
  - Da Nang Stroke Center, Da Nang
  - 115 PEOPLE's HOSPITAL, Ho Chi Minh City
  - University Medical Center, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 60 days

REFERENCES:
- [Background] Yoshimura S, Sakai N, Yamagami H, Uchida K, Beppu M, Toyoda K, Matsumaru Y, Matsumoto Y, Kimura K, Takeuchi M, Yazawa Y, Kimura N, Shigeta K, Imamura H, Suzuki I, Enomoto Y, Tokunaga S, Morita K, Sakakibara F, Kinjo N, Saito T, Ishikura R, Inoue M, Morimoto T. Endovascular Therapy for Acute Stroke with a Large Ischemic Region. N Engl J Med. 2022 Apr 7;386(14):1303-1313. doi: 10.1056/NEJMoa2118191. Epub 2022 Feb 9. PMID 35138767
- [Background] Sarraj A, Hassan AE, Abraham MG, Ortega-Gutierrez S, Kasner SE, Hussain MS, Chen M, Blackburn S, Sitton CW, Churilov L, Sundararajan S, Hu YC, Herial NA, Jabbour P, Gibson D, Wallace AN, Arenillas JF, Tsai JP, Budzik RF, Hicks WJ, Kozak O, Yan B, Cordato DJ, Manning NW, Parsons MW, Hanel RA, Aghaebrahim AN, Wu TY, Cardona-Portela P, Perez de la Ossa N, Schaafsma JD, Blasco J, Sangha N, Warach S, Gandhi CD, Kleinig TJ, Sahlein D, Elijovich L, Tekle W, Samaniego EA, Maali L, Abdulrazzak MA, Psychogios MN, Shuaib A, Pujara DK, Shaker F, Johns H, Sharma G, Yogendrakumar V, Ng FC, Rahbar MH, Cai C, Lavori P, Hamilton S, Nguyen T, Fifi JT, Davis S, Wechsler L, Pereira VM, Lansberg MG, Hill MD, Grotta JC, Ribo M, Campbell BC, Albers GW; SELECT2 Investigators. Trial of Endovascular Thrombectomy for Large Ischemic Strokes. N Engl J Med. 2023 Apr 6;388(14):1259-1271. doi: 10.1056/NEJMoa2214403. Epub 2023 Feb 10. PMID 36762865
- [Result] Huo X, Ma G, Tong X, Zhang X, Pan Y, Nguyen TN, Yuan G, Han H, Chen W, Wei M, Zhang J, Zhou Z, Yao X, Wang G, Song W, Cai X, Nan G, Li D, Wang AY, Ling W, Cai C, Wen C, Wang E, Zhang L, Jiang C, Liu Y, Liao G, Chen X, Li T, Liu S, Li J, Gao F, Ma N, Mo D, Song L, Sun X, Li X, Deng Y, Luo G, Lv M, He H, Liu A, Zhang J, Mu S, Liu L, Jing J, Nie X, Ding Z, Du W, Zhao X, Yang P, Liu L, Wang Y, Liebeskind DS, Pereira VM, Ren Z, Wang Y, Miao Z; ANGEL-ASPECT Investigators. Trial of Endovascular Therapy for Acute Ischemic Stroke with Large Infarct. N Engl J Med. 2023 Apr 6;388(14):1272-1283. doi: 10.1056/NEJMoa2213379. Epub 2023 Feb 10. PMID 36762852
- [Derived] Le TQ, Nguyen SVD, Tran TV, Pham TP, Le NV, Nguyen DT, Nguyen HH, Pham HVN, Ngo TK, Nguyen TQ, Pham TN, Cao HV, Huynh VT, Duong HQ, Chen CH, Nguyen TT. Large Core Thrombectomy: Feasibility of Simplified Protocol in Resource-Limited Settings. Stroke Vasc Interv Neurol. 2025 Sep 23;5(6):e001810. doi: 10.1161/SVIN.125.001810. eCollection 2025 Nov. PMID 41608713